CLINICAL TRIAL: NCT01200290
Title: An Exploratory/Proof of Concept Investigation of the Safety and Pharmacodynamics of LY2127399 in HLA-Presensitized Patients With End-Stage Renal Disease Awaiting Transplantation
Brief Title: A Study in Participants With End-Stage Renal Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13710; H9B-MC-BCDR (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-09-03; First posted 2010-09-13 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Kidney Failure, Chronic
Keywords: end stage renal disease; end stage kidney disease; ESRD; Uremia; Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Uremia | interventions — tabalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2127399 (Experimental)
  Interventions: Drug: LY2127399

INTERVENTIONS:
Drug: LY2127399 — 120 milligrams (mg) administered subcutaneously every 4 weeks for 20 weeks. A loading dose of 240 mg will be given as the first dose of the study medication

SUMMARY:
The purpose of this trial is to explore the effect of LY2127399 on those antibodies that are a barrier to kidney transplant. Transplantation is currently the definitive treatment for End-Stage Renal Disease (ESRD), providing prolonged survival and improved quality of life.

DETAILED DESCRIPTION:
In this study, LY2127399 will be tested as a potential treatment to reduce the blood proteins in some participants with ESRD. These proteins are called alloantibodies and are made by the body to react with other proteins on cells of transplanted organs called human leukocyte antigen (HLA) proteins. When a participant has these antibodies, they are referred to as HLA-presensitized. Often the presence of these antibodies, categorized by a method called the panel reactive antibody (PRA), can make a person ineligible to receive a transplant or experience very long wait times on the kidney transplant waiting list. Therefore the need to reduce the antibodies is significant for the successful treatment of ESRD. This study will treat ESRD participants for 6 months with LY2127399 and measure PRA levels for a total of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Have ESRD and are awaiting kidney transplant
* Have a stable PRA score >50%

Exclusion Criteria:

* Have had a tonsillectomy
* Have a semi-permanent/tunneled catheter
* Have had intravenous immunoglobulin (IVIg) in the past 6 months
* Have had plasmapheresis in the past 6 months
* Uncontrolled hypertension
* Presence of clinically significant cardiac disease in the past 6 months
* Malignancy in the past 5 years, with the exception of cervical, basal cell and squamous epithelial cell cancers
* Have active or recent infection including herpes zoster or herpes simplex in the last 30 days
* Have evidence or suspicion of active Tuberculosis (TB)
* Have had major surgery in the past 2 months
* Have had a serious infection with recovery in the past 3 months
* Have Hepatitis B or C or have Human Immunodeficiency Virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Mujtaba MA, Komocsar WJ, Nantz E, Samaniego MD, Henson SL, Hague JA, Lobashevsky AL, Higgins NG, Czader M, Book BK, Anderson MD, Pescovitz MD, Taber TE. Effect of Treatment With Tabalumab, a B Cell-Activating Factor Inhibitor, on Highly Sensitized Patients With End-Stage Renal Disease Awaiting Transplantation. Am J Transplant. 2016 Apr;16(4):1266-75. doi: 10.1111/ajt.13557. Epub 2016 Jan 18. PMID 26780484

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 24-week treatment period (Weeks 0-24) and a follow-up period (up to Week 76). Participants who discontinued study drug administration were placed into the post-treatment follow-up period.
Groups:
- LY2127399: LY2127399 was administered as a loading dose of 240-milligram (mg) subcutaneous (SC) injection at Week 0 followed by maintenance doses of 120-mg SC injections every 4 weeks at Weeks 4, 8, 12, 16 and 20.
Period: Treatment Period
Arm/Group | LY2127399
Started | 18
Received at Least 1 Dose of Study Drug | 18
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1
Period: Post-Treatment Follow-Up Period
Arm/Group | LY2127399
Started | 18 (Participant who discontinued treatment was included in the post-treatment follow-up period.)
Completed | 16
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- LY2127399: LY2127399 was administered as a loading dose of 240-mg SC injection at Week 0 followed by maintenance doses of 120-mg SC injections every 4 weeks at Weeks 4, 8, 12, 16 and 20.
Arm/Group | LY2127399
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Panel Reactive Antibodies (PRA) [Mean (Standard Deviation); unit: percentage of population] — The PRA value is calculated and expressed as a percentage, which can range from 0 percent (%) to 100%. The value represents a summation of the total HLA antibody burden that the participant has and how frequently those HLA antigens appear in organ donor population. A calculated PRA of 20% means the participant has antibodies that represent an antigen frequency that exists in approximately 20% of the population.
  percentage of population | 93.111 (10.593)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PRA
Description: The PRA value is calculated and expressed as a percentage, which can range from 0 % to 100%. The value represents a summation of the total HLA antibody burden that the participant has and how frequently those HLA antigens appear in organ donor population. A calculated PRA of 20% means the participant has antibodies that represent an antigen frequency that exists in approximately 20% of the population.
Time Frame: Baseline, Weeks 8, 16, 24, 36, 52, 64 and 76
Population: All enrolled participants who received at least 1 dose of study drug, had a non-missing baseline PRA score and at least 1 non-missing post-baseline PRA score.
Measure: Mean (Standard Deviation); unit: percentage of population
Arm/Group | LY2127399
Number analyzed (Participants) | 18
percentage of population
  Week 8 | -0.706 (2.664)
  Week 16 | -2.176 (3.575)
  Week 24 | -1.688 (3.240)
  Week 36 | -2.353 (3.499)
  Week 52 | -0.529 (3.573)
  Week 64 | -1.706 (4.497)
  Week 76 | -2.800 (7.674)
Statistical Analysis 1: Comparison: LY2127399; Test type: Superiority or Other; p = 0.324, Mixed Effect Model Repeat Measurement — P-value is for Week 8
Statistical Analysis 2: Comparison: LY2127399; Test type: Superiority or Other; p = 0.031, Mixed Effect Model Repeat Measurement — P-value is for Week 16
Statistical Analysis 3: Comparison: LY2127399; Test type: Superiority or Other; p = 0.076, Mixed Effect Model Repeat Measurement — P-value is for Week 24
Statistical Analysis 4: Comparison: LY2127399; Test type: Superiority or Other; p = 0.013, Mixed Effect Model Repeat Measurement — P-value is for Week 36
Statistical Analysis 5: Comparison: LY2127399; Test type: Superiority or Other; p = 0.553, Mixed Effect Model Repeat Measurement — P-value is for Week 52
Statistical Analysis 6: Comparison: LY2127399; Test type: Superiority or Other; p = 0.132, Mixed Effect Model Repeat Measurement — P-value is for Week 64
Statistical Analysis 7: Comparison: LY2127399; Test type: Superiority or Other; p = 0.230, Mixed Effect Model Repeat Measurement — P-value is for Week 76

2. Primary Outcome: Change From Baseline in Arcsine Transformed PRA Scores
Description: The PRA value is calculated and expressed as a percentage, which can range from 0% to 100%. The value represents a summation of the total HLA antibody burden that the participant has and how frequently those HLA antigens appear in organ donor population. A calculated PRA of 20% means the participant has antibodies that represent an antigen frequency that exists in approximately 20% of the population. PRA scores were transformed using the arcsine function, which enables a skewed distribution of data typically expressed as proportions to achieve properties closer to a normal distribution. The range of possible arcsine transformed PRA scores is 0 (when PRA = 0) to approximately 1.57 (when PRA =100). Higher scores indicate the participant has antibodies against HLA antigens that appear frequently in the organ donor population.
Time Frame: Baseline, Weeks 8, 16, 24, 36, 52, 64 and 76
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399
Number analyzed (Participants) | 18
units on a scale
  Week 8 | -0.022 (0.086)
  Week 16 | -0.059 (0.101)
  Week 24 | -0.060 (0.104)
  Week 36 | -0.078 (0.099)
  Week 52 | -0.014 (0.133)
  Week 64 | -0.053 (0.124)
  Week 76 | -0.071 (0.158)
Statistical Analysis 1: Comparison: LY2127399; Test type: Superiority or Other; p = 0.335, Mixed Effect Model Repeat Measurement — P-value is for Week 8
Statistical Analysis 2: Comparison: LY2127399; Test type: Superiority or Other; p = 0.043, Mixed Effect Model Repeat Measurement — P-value is for Week 16
Statistical Analysis 3: Comparison: LY2127399; Test type: Superiority or Other; p = 0.073, Mixed Effect Model Repeat Measurement — P-value is for Week 24
Statistical Analysis 4: Comparison: LY2127399; Test type: Superiority or Other; p = 0.004, Mixed Effect Model Repeat Measurement — P-value is for Week 36
Statistical Analysis 5: Comparison: LY2127399; Test type: Superiority or Other; p = 0.699, Mixed Effect Model Repeat Measurement — P-value is for Week 52
Statistical Analysis 6: Comparison: LY2127399; Test type: Superiority or Other; p = 0.095, Mixed Effect Model Repeat Measurement — P-value is for Week 64
Statistical Analysis 7: Comparison: LY2127399; Test type: Superiority or Other; p = 0.082, Mixed Effect Model Repeat Measurement — P-value is for Week 76

3. Secondary Outcome: Change From Baseline in Serum Immunoglobulin Levels
Description: Immunoglobulins (Ig), or antibodies, are large molecular weight proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Change from baseline in serum immunoglobulin A (IgA), immunoglobulin G (IgG), IgG1-4, and immunoglobulin M (IgM) levels are reported. A negative change indicates a decrease in Ig levels.
Time Frame: Baseline, Weeks 8, 16, 24, 36 and 52
Population: All enrolled participants who received at least 1 dose of study drug, had a non-missing baseline Ig value and at least 1 non-missing post-baseline Ig value.
Measure: Mean (Standard Deviation); unit: grams/liter (g/L)
Arm/Group | LY2127399
Number analyzed (Participants) | 18
grams/liter (g/L)
  IgA at Week 8 | -0.305 (0.4552)
  IgA at Week 16 | -0.261 (0.3983)
  IgA at Week 24 | -0.409 (0.5467)
  IgA at Week 36 | -0.325 (0.5715)
  IgA at Week 52 | -0.098 (0.5090)
  IgG at Week 8 | -1.625 (1.8500)
  IgG at Week 16 | -1.856 (1.5373)
  IgG at Week 24 | -2.048 (1.8486)
  IgG at Week 36 | -2.245 (2.1388)
  IgG at Week 52 | -0.625 (3.0933)
  IgG1 at Week 8 | -1.018 (1.4024)
  IgG1 at Week 16 | -1.459 (1.5242)
  IgG1 at Week 24 | -1.682 (1.8190)
  IgG1 at Week 36 | -1.969 (1.6652)
  IgG1 at Week 52 | -0.668 (2.9531)
  IgG2 at Week 8 | -0.125 (0.3016)
  IgG2 at Week 16 | -0.261 (0.3044)
  IgG2 at Week 24 | -0.274 (0.2693)
  IgG2 at Week 36 | -0.226 (0.3951)
  IgG2 at Week 52 | 0.046 (0.5918)
  IgG3 at Week 8 | -0.046 (0.0847)
  IgG3 at Week 16 | -0.072 (0.0601)
  IgG3 at Week 24 | -0.076 (0.0899)
  IgG3 at Week 36 | -0.061 (0.1074)
  IgG3 at Week 52 | -0.022 (0.0761)
  IgG4 at Week 8 | 0.013 (0.0511)
  IgG4 at Week 16 | -0.009 (0.0512)
  IgG4 at Week 24 | -0.010 (0.0500)
  IgG4 at Week 36 | -0.032 (0.0558)
  IgG4 at Week 52 | 0.019 (0.0899)
  IgM at Week 8 | -0.208 (0.2650)
  IgM at Week 16 | -0.295 (0.2895)
  IgM at Week 24 | -0.266 (0.2781)
  IgM at Week 36 | -0.302 (0.2449)
  IgM at Week 52 | -0.197 (0.3032)

4. Secondary Outcome: Percent Change From Baseline at Week 1 and Week 24 in Relative Percent of Lymphocytes for B Cell Populations in the Tonsil
Description: B cell population counts are: Total B cells [cluster designation (CD)19+], mature naïve B cells [CD19+CD27-immunoglobulin D (IgD)+CD10-], switched memory B cells (CD19+CD27+IgD-), unswitched memory B cells (CD19+CD27+IgD+), germinal center B cells Bm2&apos (CD19+CD38+IgD+), germinal center B cells Bm3, Bm4 (CD19+CD38+IgD-), germinal center B cells (CD19+CD38+CD10+CD71+), transitional (Tr) B cells (CD19+CD38++/+++CD24+++/+CD10+) and Tr B cells (CD19+CD27-IgD+CD10+).
Time Frame: Baseline, Weeks 1 and 24
Population: All enrolled participants who received at least 1 dose of study drug, had a non-missing baseline tonsil B cell populations value and at least 1 non-missing post-baseline B cell populations value.
Measure: Mean (Standard Deviation); unit: relative percent of Lymphocytes
Arm/Group | LY2127399
Number analyzed (Participants) | 10
relative percent of Lymphocytes
  Total B cells at Week 1 | 12.732 (61.2266)
  Total B cells at Week 24 | -25.371 (40.1642)
  Mature naïve at Week 1 | -1.559 (4.9348)
  Mature naïve at Week 24 | -21.611 (12.6669)
  Switched memory at Week 1 | 11.850 (27.6106)
  Switched memory at Week 24 | 92.905 (74.1293)
  Unswitched memory at Week 1 | 40.343 (82.3486)
  Unswitched memory at Week 24 | 224.298 (331.6551)
  Germinal center Bm2' at Week 1 | -8.818 (21.9800)
  Germinal center Bm2' at Week 24 | -61.051 (20.9845)
  Germinal center Bm3, Bm4 at Week 1 | 26.705 (51.6762)
  Germinal center Bm3, Bm4 at Week 24 | 104.890 (230.9829)
  Germinal center at Week 1 | 7.280 (58.0681)
  Germinal center at Week 24 | 19.279 (102.9617)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 1 | 46.508 (96.0036)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 24 | 26.999 (79.5306)
  Tr (CD19+CD27-IgD+CD10+) at Week 1 | -8.977 (53.7335)
  Tr (CD19+CD27-IgD+CD10+) at Week24 | -59.131 (27.2120)

5. Secondary Outcome: Percent Change From Baseline in Relative Percent of Lymphocytes for B Cell Populations in Peripheral Blood
Description: B cell population counts are: Total B cells (CD19+), mature naïve B cells (CD19+CD27-IgD+CD10-), switched memory B cells (CD19+CD27+IgD-), unswitched memory B cells (CD19+CD27+IgD+), Tr B cells (CD19+CD38++/+++CD24+++/+CD10+) and Tr B cells (CD19+CD27-IgD+CD10+).
Time Frame: Baseline, Weeks1, 4, 8, 16, 24, 36, 52, 64 and 76
Population: All enrolled participants who received at least 1 dose of study drug, had a non-missing baseline peripheral blood B cell populations value and at least 1 non-missing post-baseline B cell populations value.
Measure: Mean (Standard Deviation); unit: relative percent of Lymphocytes
Arm/Group | LY2127399
Number analyzed (Participants) | 18
relative percent of Lymphocytes
  Total B cells at Week 1 | 35.303 (34.2864)
  Total B cells at Week 4 | -10.883 (24.1837)
  Total B cells at Week 8 | -28.765 (25.2472)
  Total B cells at Week 16 | -45.027 (23.1939)
  Total B cells at Week 24 | -52.115 (22.5144)
  Total B cells at Week 36 | -63.677 (17.2158)
  Total B cells at Week 52 | -60.808 (17.8105)
  Total B cells at Week 64 | -25.982 (49.3294)
  Total B cells at Week 76 | -32.467 (32.7608)
  Mature naïve at Week 1 | -1.172 (11.6626)
  Mature naïve at Week 4 | -14.222 (13.8931)
  Mature naïve at Week 8 | -34.496 (15.9776)
  Mature naïve at Week 16 | -47.957 (19.0080)
  Mature naïve at Week 24 | -54.859 (23.8066)
  Mature naïve at Week 36 | -54.030 (20.4375)
  Mature naïve at Week 52 | -20.440 (29.5837)
  Mature naïve at Week 64 | -1.237 (22.1831)
  Mature naïve at Week 76 | 9.210 (21.7629)
  Switched memory at Week 1 | 20.241 (41.7855)
  Switched memory at Week 4 | 111.611 (73.4853)
  Switched memory at Week 8 | 204.443 (118.2768)
  Switched memory at Week 16 | 305.653 (198.0679)
  Switched memory at Week 24 | 305.930 (197.4446)
  Switched memory at Week 36 | 285.668 (238.3301)
  Switched memory at Week 52 | 75.155 (85.9638)
  Switched memory at Week 64 | 20.179 (42.5419)
  Switched memory at Week 76 | 11.947 (37.6837)
  Unswitched memory at Week 1 | 5.563 (41.2351)
  Unswitched memory at Week 4 | 45.073 (61.3175)
  Unswitched memory at Week 8 | 110.285 (87.0203)
  Unswitched memory at Week 16 | 143.020 (113.1325)
  Unswitched memory at Week 24 | 138.646 (121.7276)
  Unswitched memory at Week 36 | 140.917 (123.0888)
  Unswitched memory at Week 52 | 65.607 (109.5101)
  Unswitched memory at Week 64 | 17.782 (41.1260)
  Unswitched memory at Week 76 | 26.283 (52.1802)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 1 | -13.511 (29.4311)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 4 | -49.869 (23.7764)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 8 | -49.292 (18.5600)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 16 | -40.847 (36.9400)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 24 | -44.355 (32.0001)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 36 | 10.080 (118.1582)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 52 | 36.776 (136.3827)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 64 | 9.357 (210.4455)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 76 | -7.396 (181.0879)
  Tr (CD19+CD27-IgD+CD10+) at Week1 | -6.512 (23.6020)
  Tr (CD19+CD27-IgD+CD10+) at Week4 | -42.852 (25.4319)
  Tr (CD19+CD27-IgD+CD10+) at Week8 | -56.047 (13.9734)
  Tr (CD19+CD27-IgD+CD10+) at Week 16 | -56.886 (32.9379)
  Tr (CD19+CD27-IgD+CD10+) at Week 24 | -64.706 (24.3874)
  Tr (CD19+CD27-IgD+CD10+) at Week 36 | -41.231 (48.6871)
  Tr (CD19+CD27-IgD+CD10+) at Week 52 | 6.504 (118.6276)
  Tr (CD19+CD27-IgD+CD10+) at Week 64 | 2.059 (177.4749)
  Tr (CD19+CD27-IgD+CD10+) at Week 76 | -45.425 (90.9992)

6. Secondary Outcome: Percent Change From Baseline in Absolute Counts of B Cell Populations in Peripheral Blood
Description: as for outcome 5
Time Frame: Baseline, Weeks1, 4, 8, 16, 24, 36 and 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change in absolute counts
Arm/Group | LY2127399
Number analyzed (Participants) | 18
percent change in absolute counts
  Total B cells at Week 1 | 37.305 (48.2410)
  Total B cells at Week 4 | -12.050 (48.5995)
  Total B cells at Week 8 | -27.875 (51.5586)
  Total B cells at Week 16 | -46.861 (33.8978)
  Total B cells at Week 24 | -55.759 (33.6090)
  Total B cells at Week 36 | -68.301 (23.1588)
  Total B cells at Week 52 | -65.676 (17.3689)
  Mature naïve at Week 1 | 37.533 (60.6785)
  Mature naïve at Week 4 | -23.351 (47.2486)
  Mature naïve at Week 8 | -52.128 (39.7386)
  Mature naïve at Week 16 | -72.891 (19.8886)
  Mature naïve at Week 24 | -81.367 (16.4389)
  Mature naïve at Week 36 | -85.213 (12.9636)
  Mature naïve at Week 52 | -70.114 (21.6407)
  Switched memory at Week 1 | 64.309 (68.7102)
  Switched memory at Week 4 | 66.849 (62.1042)
  Switched memory at Week 8 | 83.774 (76.5159)
  Switched memory at Week 16 | 74.667 (72.0109)
  Switched memory at Week 24 | 56.192 (117.0402)
  Switched memory at Week 36 | 1.221 (53.8382)
  Switched memory at Week 52 | -48.620 (17.2563)
  Unswitched memory at Week 1 | 51.590 (98.1357)
  Unswitched memory at Week 4 | 17.522 (62.0773)
  Unswitched memory at Week 8 | 35.339 (84.7680)
  Unswitched memory at Week 16 | 11.962 (74.5105)
  Unswitched memory at Week 24 | -8.604 (59.8587)
  Unswitched memory at Week 36 | -33.746 (38.8791)
  Unswitched memory at Week 52 | -48.381 (26.9717)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 1 | 22.103 (72.4137)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 4 | -57.052 (30.7060)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 8 | -64.282 (25.8516)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 16 | -71.138 (26.0579)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 24 | -80.746 (12.1379)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 36 | -75.133 (20.0926)
  Tr(CD19+CD38++/+++CD24+++/+CD10+) at Week 52 | -59.288 (31.9767)
  Tr(CD19+CD27-IgD+CD10+) at Week 1 | 25.018 (44.8425)
  Tr(CD19+CD27-IgD+CD10+) at Week 4 | -47.991 (42.3991)
  Tr(CD19+CD27-IgD+CD10+) at Week 8 | -70.447 (20.1950)
  Tr(CD19+CD27-IgD+CD10+) at Week 16 | -76.085 (24.0089)
  Tr(CD19+CD27-IgD+CD10+) at Week 24 | -87.204 (11.6008)
  Tr(CD19+CD27-IgD+CD10+) at Week 36 | -84.531 (14.5977)
  Tr(CD19+CD27-IgD+CD10+) at Week 52 | -69.306 (29.8739)

7. Secondary Outcome: Population Pharmacokinetics (PK): Constant Clearance
Description: Population estimate of constant clearance as determined by population PK analysis. A 2-compartment model was used in PK modeling. Constant clearance is the PK parameter which describes the linear elimination of LY2127399 from serum.
Time Frame: Baseline through Week 24
Population: All randomized participants who received at least 1 dose of LY2127399 with evaluable LY2127399 PK data.
Measure: Mean (Standard Error); unit: milliliters/hour (mL/h)
Arm/Group | LY2127399
Number analyzed (Participants) | 18
milliliters/hour (mL/h) | 5.65 (9.72)

8. Primary Outcome: Number of Participants With a Change From Baseline Positive to Post-Baseline Negative in the Summation of Top 10 Highest Antibody Levels (Class I and Class II Single Antigen Reactivity Reported Separately) During Treatment and Follow-Up
Time Frame: Baseline through Weeks 24, 52 and 76
Population: All enrolled participants who received at least 1 dose of study drug and had single antigen reactivity assessed at baseline, during treatment and during follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2127399
Number analyzed (Participants) | 18
Participants
  Class I - Week 24 | 0
  Class I - Week 52 | 0
  Class I - Week 76 | 0
  Class II - Week 24 | 0
  Class II - Week 52 | 0
  Class II - Week 76 | 0

ADVERSE EVENTS:
Arm/Group | LY2127399
Serious Adverse Events (participants affected / at risk) | 9/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2127399 (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2127399 (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 2 (2)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Catheter site pain (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Feeling abnormal (General disorders) | 1 (1)
Injection site extravasation (General disorders) | 2 (3)
Injection site pain (General disorders) | 17 (83)
Medical device complication (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (5)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 3 (3)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Cardiac murmur (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Uraemic neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Communication disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1)
Uterine cyst (Reproductive system and breast disorders) | 1/10 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 5 (7)
Iliac vein occlusion (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days